CLINICAL TRIAL: NCT05722574
Title: Project Relate: Romantic Relationship Competence Single-Session Intervention Trial
Brief Title: Project Relate: Romantic Relationship Competence SSI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Jessica Schleider, Assistant Professor, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB2022-00262
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Relational Problems; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either the intervention condition or the information-only control group.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Information Only Control Condition (Active Comparator): The information only control condition is designed to mimic relationship education that could be easily found online by adolescents. This condition does not teach romantic competence skills such as insight, communication/mutuality, or emotion regulation skills; rather, it focuses on educating subjects about the healthy and unhealthy signs of a romantic relationship. In addition, this condition is designed to control for nonspecific aspects of the intervention, such as engaging in an online program and taking time to reflect on one's relationships.
  Interventions: Behavioral: Information Only Control Condition
- Romantic Competence Intervention (Experimental): The Romantic Competence Single-Session Intervention provides adolescents with the opportunity to learn one of three relational skills online: (1) Insight, the ability to understand what one needs in relationships and act in alignment with one's needs, (2) Communication, the capacity to listen to others and express one's needs effectively, and (3) Stay vs. Go, the ability to reflect and make difficult decisions in relationships. Adolescents are presented with the opportunity to choose which module they would like to complete. Each module has the following components: psychoeducation, a personalized action plan, and practice overcoming barriers.
  Interventions: Behavioral: Romantic Competence Intervention

INTERVENTIONS:
Behavioral: Romantic Competence Intervention — Online, 30-minute self-administered relationship competence program for youth ages 16-20
  Arms: Romantic Competence Intervention
Behavioral: Information Only Control Condition — Online, 30-minute self-administered relationship education activity for youth ages 16-20
  Arms: Information Only Control Condition

SUMMARY:
The COVID-19 pandemic has increased social isolation and depressive symptoms in youth, adding strain to an already overwhelmed mental healthcare system. Online single-session interventions are digital programs that can help expand access to care and teach evidence-based skills. To help youth build healthy relationships, we developed 3 online single-session interventions (SSI) to teach romantic competence skills to adolescents and emerging adults. Youth, ages 16-20, will be recruited to social media and randomly assigned to one of two conditions: the intervention condition, offering them three SSIs to select from, or an information-only control group. Within the intervention condition, youth will complete one of three romantic competence SSIs: (1) Insight, targeting awareness of one's needs in relationships, (2) Communication, teaching listening and communication skills, and (3) Stay vs. Go, helping youth make difficult decisions. Investigators will assess each SSI's relative benefits on relationship knowledge and depressive symptoms up to three months later compared to the information-only control group. Results will reveal if online SSIs can teach romantic competence skills and if engaging in these interventions has psychosocial benefits for youth with elevated depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* are fluent in English
* have consistent internet and computer/laptop/smartphone access
* report elevated depressive symptoms (a score of >2 on the Patient Health Questionnaire-2 item version [PHQ-2])

Exclusion Criteria:

* fail to meet the above-listed inclusion criteria
* exit the study prior to condition randomization
* respond with either copy/pasted responses from text earlier in the intervention to any of free response questions
* obvious lack of English fluency in open response questions
* responding with random text in open response questions
* duplicate responses from the same individual in baseline or follow-up surveys

Ages: 16 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9; Kroenke et al., 2001) | Pre-SSI to 3-month follow-up
  The PHQ-9 is a reliable, valid measure of depression symptom severity. Higher scores indicate more severe symptoms of depression.

SECONDARY OUTCOMES:
Beck Hopelessness Scale - 4 Item Version (Steed, 2001) | Pre-Intervention to Immediately Post-Intervention; Pre-Intervention to 3-month follow-up
  This scale asks participants to rate 4 statements based on their sense of hopelessness. Participants rate the 4 statements on a 4 point scale ranging from 0 (Absolutely Disagree) to 3 (Absolutely Agree). Average scores across all items range from 0 to 3, with a higher score indicating greater levels of hopelessness.
Relationship Learning Inventory (Davila et al., 2000) | Pre-Intervention to Immediately Post-Intervention
  This measure uses 3 questions post-intervention to assess the extent to which participants gained learned something important after the activity, thought about relationships differently, or felt validated in the way that they have been thinking/acting in their relationships.
Generalized Anxiety Disorder (GAD-7; Steed, 2001) | Pre-SSI to 3-month follow-up
  The GAD-7 measures the severity of clinical anxiety symptoms, based on diagnostic criteria for generalized anxiety disorder. The GAD-7 includes 7 items asking respondents how often, during the last 2 weeks, they were bothered by each of 7 anxiety symptoms. Higher scores reflect higher generalized anxiety symptoms.
Relationship Decision Making Scale (Vennum & Fincham, 2011) | Pre-SSI to 3-month follow-up
  The Relationship Deciding Scale measures effective decision-making during interpersonal situations. It has three subscales with items rated on a 5- point scale (1 = strongly disagree, 5 = strongly agree), relationship confidence, assessing confidence in maintaining a relationship; warning signs, assessing awareness of and ability to deal with warning signs in relationships; and deciding, assessing thoughtfulness regarding decisions. Higher scores suggest more effective decision-making.
Relationship Knowledge and Efficacy Scale (Davila et al., 2020) | Pre-SSI to 3-month follow-up
  This measure consists of 21 items, rated 1-7 (1 = strongly disagree, 7 = strongly agree), and measures six domains: (1) confidence in one's knowledge about what a healthy relationship is and ability to manage relationships; (2) confidence in one's knowledge about and ability to cope with relationship problems; (3) willingness to compromise oneself; (4) beliefs that any relationship can work if you work hard enough; and (5) overreliance on emotions for relationship decisions. Higher scores reflect better relationship knowledge and efficacy.
Qualitative Changes in the Relationship Learning Inventory | Immediately Post-Intervention
  Immediately after the activity, participants will be asked, "In your opinion, what was the most important thing you learned from this activity?" "Based on what you learned, will you do anything differently in your relationships? If yes, please elaborate on what you will do differently." At the 3-month follow-up, we also ask two additional questions, "From what you remember, what was the most important thing you learned in our relationship education activity?" and "Since completing this activity, have you noticed any changes in how you navigate your relationships? If yes, please tell us what you have noticed." Participants are provided with space to answer these questions via text entry.

OTHER OUTCOMES:
UCLA Loneliness Scale | Pre-SSI to 3-month follow-up
  The ULS is a widely used self-report scale of loneliness. The brief 3-item version will be used here. Participants will rate agreement with 3 items reflecting loneliness (e.g. "I feel left out"; "I feel isolated from others"). Higher scores reflect higher levels of loneliness.
Perceived Changes | Immediately Post-Intervention
  Participants are asked 3 questions about perceived changes in mood, hopelessness, and problem-solving capabilities. "Compared to before doing this activity, to what extent are you feeling hopeless right now?" Items are rated 1-5 (1 = much more hopeless, 5 = much less hopeless).
  Compared to before doing this activity, what is your mood like right now?" Items are rated 1-5 (1 = much worse, 5 = much better).
  "Compared to before doing this activity, to what extent are you able to solve the problems facing you right now?" Items are rated 1-5 (1 = much less able to solve problems, 5 = a lot more able to solve problems).
Program Feedback Scale | Pre-Intervention to Immediately Post-Intervention
  The PFS asks youth to rate agreement with 7 statements indicating perceived acceptability of an SSI (e.g. "I enjoyed the program") on a 5-point Likert scale (1="really disagree"; 5="totally agree"). A score of 3.5/5 or above on any given PFS item is interpreted as an "acceptable" rating on that item. Scores are calculated at the item-level, and higher scores reflect greater acceptability for each item.
Global/General Attachment (ECR-RS, 9-item Version; Fraley et al., 2015) | Pre-SSI to 3-month follow-up
  The Relationship Structures Questionnaire is a self-report measure that assesses general attachment patterns across a variety of close relationships. It asks participants to rate the extent to which each statement describes their feelings about close relationships in general. This abbreviated measure consists of 9 items, ranking from 1 (Strongly Disagree) to 7 (Strongly Agree). This measure consists of two subscales: anxiety and avoidance. Higher scores on the anxiety and avoidance subscales represent higher levels of attachment insecurity.
Interpersonal Reactivity Index (Peloquin & Lafontaine, 2010). | Pre-SSI to 3-month follow-up
  We assessed empathy and perspective-taking with the two subscales of the Interpersonal Reactivity Index (IRIC; Péloquin & Lafontaine; 2010); this measure was only administered to youth who were dating or in a committed romantic relationship. Items rated on a 5-point scale (0 = does not describe me well, 4 = describes me very well). Example items for perspective taking include, "When I'm upset at my partner, I usually try to 'put myself in his/her shoes' for a while" and empathic concern, " I often have tender, concerned feelings for my partner when he/she is less fortunate than me." Participants were instructed to 'Answer about your current or most recent partner,' and higher scores reflect higher levels of empathy and perspective-taking, respectively.
Couple Satisfaction Index (CSI-4; Funk & Rogge, 2007). | Pre-SSI to 3-month follow-up
  We used the 4-item measure from the Couple Satisfaction Index to measure relationship satisfaction; this measure was administered to youth who were dating or in a committed romantic relationship. Items include questions like "How rewarding is your relationship with your partner?" and "In general, how satisfied are you with your relationship?" Items are ranked 0- Not at all to 5- Completely. CSI-4 scores can range from 0 to 21. Higher scores indicate higher levels of relationship satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Schleider, PhD, Principal Investigator — Stony Brook University

IPD SHARING:
Plan to Share IPD: Yes
After our trial has ended, data without any identifying markers will be made available to researchers interested in our dataset.
Supporting Information: Study Protocol, SAP
Time Frame: Deidentified data will be made available on the Open Science Framework within one year of publishing study results.
Access Criteria: Access will not be restricted.

REFERENCES:
- [Background] Avenevoli S, Swendsen J, He JP, Burstein M, Merikangas KR. Major depression in the national comorbidity survey-adolescent supplement: prevalence, correlates, and treatment. J Am Acad Child Adolesc Psychiatry. 2015 Jan;54(1):37-44.e2. doi: 10.1016/j.jaac.2014.10.010. Epub 2014 Oct 29. PMID 25524788
- [Background] Marques de Miranda D, da Silva Athanasio B, Sena Oliveira AC, Simoes-E-Silva AC. How is COVID-19 pandemic impacting mental health of children and adolescents? Int J Disaster Risk Reduct. 2020 Dec;51:101845. doi: 10.1016/j.ijdrr.2020.101845. Epub 2020 Sep 10. PMID 32929399
- [Background] Schleider JL, Weisz JR. Little Treatments, Promising Effects? Meta-Analysis of Single-Session Interventions for Youth Psychiatric Problems. J Am Acad Child Adolesc Psychiatry. 2017 Feb;56(2):107-115. doi: 10.1016/j.jaac.2016.11.007. Epub 2016 Nov 25. PMID 28117056
- [Background] Osborn TL, Rodriguez M, Wasil AR, Venturo-Conerly KE, Gan J, Alemu RG, Roe E, Arango G S, Otieno BH, Wasanga CM, Shingleton R, Weisz JR. Single-session digital intervention for adolescent depression, anxiety, and well-being: Outcomes of a randomized controlled trial with Kenyan adolescents. J Consult Clin Psychol. 2020 Jul;88(7):657-668. doi: 10.1037/ccp0000505. Epub 2020 May 11. PMID 32391709
- [Background] Schleider JL, Mullarkey MC, Fox KR, Dobias ML, Shroff A, Hart EA, Roulston CA. A randomized trial of online single-session interventions for adolescent depression during COVID-19. Nat Hum Behav. 2022 Feb;6(2):258-268. doi: 10.1038/s41562-021-01235-0. Epub 2021 Dec 9. PMID 34887544
- [Background] Pilkonis PA, Choi SW, Reise SP, Stover AM, Riley WT, Cella D; PROMIS Cooperative Group. Item banks for measuring emotional distress from the Patient-Reported Outcomes Measurement Information System (PROMIS(R)): depression, anxiety, and anger. Assessment. 2011 Sep;18(3):263-83. doi: 10.1177/1073191111411667. Epub 2011 Jun 21. PMID 21697139
- [Background] Zhang WC, Jia CX, Hu X, Qiu HM, Liu XC. Beck Hopelessness Scale: Psychometric Properties Among Rural Chinese Suicide Attempters and Non-Attempters. Death Stud. 2015;39(7):442-6. doi: 10.1080/07481187.2014.970300. Epub 2015 Feb 13. PMID 25679324
- [Background] Ahlen J, Ghaderi A. Evaluation of the Children's Depression Inventory-Short Version (CDI-S). Psychol Assess. 2017 Sep;29(9):1157-1166. doi: 10.1037/pas0000419. Epub 2016 Dec 5. PMID 27918174
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Davila J, Zhou J, Norona J, Bhatia V, Mize L, Lashman K. Teaching romantic competence skills to emerging adults: A relationship education workshop. Pers Relatsh. 2021;28(2):251-275. doi:10.1111/pere.12366
- [Background] Davila J, Mattanah J, Bhatia V, et al. Romantic competence, healthy relationship functioning, and well-being in emerging adults. Pers Relatsh. 2017;24(1):162-184. doi:10.1111/pere.12175
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941